CLINICAL TRIAL: NCT04968470
Title: Prospective Observational Study About SEBBIN Silicone Gel-filled Testicular Implants
Brief Title: SEBBIN Silicone Gel-filled Testicular Implants
Status: Recruiting | Type: Observational
Sponsor: Groupe SEBBIN (Industry)
Responsible Party: Sponsor
Other Study IDs: PEC 19-05-001
Record Dates: First submitted 2021-07-06; First posted 2021-07-20 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Complication; Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is part of the clinical evaluation of SEBBIN silicone gel-filled testicular implants, included in the technical file of the device. The aim of the study is to gather additional data about the safety and effectiveness of the device.

ELIGIBILITY:
Inclusion Criteria:

* The patient is an adult or a child at the time of implant placement with SEBBIN implant.
* The patient is candidate to a unilateral or bilateral testicular implant placement with SEBBIN implant.
* The patient has been informed of the study, has read the patient information letter and -provided oral consent.

Exclusion Criteria:

* The patient has silicone implants somewhere else than in the scrotal sac.
* The patient was diagnosed with one of the following pathologies:

  * Systemic lupus erythematous, Sjogren syndrome, scleroderma, polymyositis, or any other connective tissue disease.
  * Rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondyloarthropathies, or any other inflammatory arthritic disease.
  * Arthritis, fibromyalgia, chronic fatigue syndrome, or any other mechanic or degenerative non-inflammatory rheumatic disease.
* The patient has a pathology that could delay healing.
* Custom-designed implants are used for surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The intended target population for the silicone gel-filled testicular implants of Groupe SEBBIN is any patient (children or adults) with agenesis or testicular atrophy, undescended testicle, testicular tumour, epididymitis / orchitis, or a trauma, for whom an orchidectomy with placement of a testicular prosthesis is indicated. Testicular implants are also indicated for sex reassignment surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Complication rate | At 10 years of follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- UZ Gent, Ghent, Belgium
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France